CLINICAL TRIAL: NCT01557387
Title: Real-time Diagnosis of Pseudopolyps During Colonoscopy Using Noninvasive Advanced Endoscopic Techniques - a Prospective Study
Brief Title: Real-time Diagnosis of Pseudopolyps During Colonoscopy
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Olympus America, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel A. Sussman, MD, MSPH, Principal Investigator, University of Miami
Other Study IDs: 20091017
Record Dates: First submitted 2011-08-11; First posted 2012-03-19 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Pseudopolyp; Inflammatory Bowel Disease
Keywords: Pseudopolyp; Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with pseudopolyps.: No treatment involved in this study.
  Interventions: Other: Endoscopic techniques

INTERVENTIONS:
Other: Endoscopic techniques — All patients will undergo non-invasive endoscopic techniques considered standard of care in surveillance for dysplasia

SUMMARY:
Significance: Biopsy of potentially benign pseudopolyps and the surrounding mucosa adds expense and prolongs the time of endoscopic procedures. Use of endoscopic technologies could decrease the need and expense of endoscopic biopsy for these lesions.

Hypothesis: Pseudopolyps will have a distinctive pattern with the specialized imaging techniques of high definition imaging, narrow band imaging, and endoscopic dye-spraying techniques using indigo carmine which will predict diagnosis without biopsy.

100 patients with inflammatory bowel disease will be enrolled in the study. Following a standard bowel preparation, each patient will be evaluated using standard endoscopic equipment. All patients will receive a standard bowel preparation (sodium phosphate, PEG-3350, or magnesium citrate based preparations). All colonoscopic evaluations will be performed for indications unrelated to the present study, including evaluation of response to medical treatment, routine surveillance exams for dysplasia, diarrhea, or rectal bleeding. Polypoid lesions will be examined using four consecutive methods: (a) high definition white light, (b) narrow band imaging, (c) chromoendoscopy (high definition white light with indigo carmine dye-spraying), and (d) histologic examination following biopsy. The flat mucosa surrounding the polypoid lesions will also be examined using theses four techniques in an effort to identify dysplastic tissue associated with these polypoid growths.

High definition white light is the standard imaging modality used for colonoscopy. Narrow band imaging (blue wavelength of light) is also used routinely and is available on all current generation colonoscopes with the press of a button. Our division routinely uses chromoendoscopy as part of surveillance for dysplasia in patients with inflammatory bowel disease. Dye spraying catheters or flushing will be utilized for dye application to mucosa. The dye used will be indigo carmine.

Directed biopsy specimens will then be performed using a multibite forceps for targeted biopsies. Routine biopsies will be performed as clinically indicated. Pathology slides will be reviewed by the gastrointestinal pathologists at the University of Miami. The gastroenterologist's interpretation based on each of the three successive endoscopic methods will then be compared to the histologic evaluation with each individual lesion serving as its own control.

DETAILED DESCRIPTION:
The colonoscopy with biopsies will be done as standard of care; additional biopsies will be taken for research purposes as detailed above. All of the imaging techniques are part of the accepted standard of care as follows: high definition white light, narrow band imaging, chromoendoscopy, and histologic examination following biopsy. Comparison of the predictive values of the imaging modalities in predicting histology from biopsy underlies the primary question of this research protocol. Cost analysis of modalities versus histology will also be performed. Time for use of the individual modalities will be recorded.

Subjects will be identified by one of the investigators during their outpatient clinic visits or while inpatient at University of Miami Hospital. Subjects who meet the inclusion/exclusion criteria and are scheduled to undergo a colonoscopy for standard of care purposes will be asked to participate in the study. Patients over 18 years of age with a confirmed diagnosis of inflammatory bowel disease with plans for routine colonoscopic evaluation and able to provide informed consent will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients equal to or over 18 years of age with a confirmed diagnosis of inflammatory bowel disease with plans for routine colonoscopic evaluation and able to provide informed consent will be included.

Exclusion Criteria:

* Patients under 18 years of age.
* Patient unwilling or unable to undergo colonoscopy with biopsies or preparation for colonoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients with inflammatory bowel disease (IBD) will be enrolled in the study. They will be identified from a population of patients undergoing colonoscopy for diagnostic purposes with IBD.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of non-invasive endoscopic techniques for diagnosis of pseudopolyps as compared to histology as the gold standard for diagnosis | 2 years or until 100 patients enrolled, whichever comes first

SECONDARY OUTCOMES:
Cost of non-invasive endoscopic techniques for diagnosis of pseudopolyps as compared to histology as the gold standard for diagnosis | 2 years or until 100 patients enrolled, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Sussman, MD, MSPH, Principal Investigator — University of Miami Division of Gastroenterology
Locations (2):
- United States (2):
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Miami Hospital, Miami, Florida

REFERENCES:
- [Derived] Sussman DA, Barkin JA, Martin AM, Varma T, Clarke J, Quintero MA, Barkin HB, Deshpande AR, Barkin JS, Abreu MT. Development of Advanced Imaging Criteria for the Endoscopic Identification of Inflammatory Polyps. Clin Transl Gastroenterol. 2015 Nov 19;6(11):e128. doi: 10.1038/ctg.2015.51. PMID 26583503